CLINICAL TRIAL: NCT07165431
Title: Clinical Evaluation of a Postbiotic Supplement in Overweight and Obese Subjects: A Randomized Controlled Trial.
Brief Title: Effect of a Postbiotic Supplementation in Overweight and Obese Subjects: A Randomized Controlled Trial (PARABIOTICS-2).
Acronym: PARABIOTICS-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARABIOTICS-2 (2025.113 Mod1)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Nutrition, Healthy; Weight Loss; Overweight and Obesity
Keywords: Postbiotic; Obesity; Nutritional advice; Microbiota; Glucose tolerance
MeSH Terms: conditions — Weight Loss; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Parallel groups, 12-week randomized nutritional intervention
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postbiotic group (Experimental): Gummy containing postbiotic formula.
  Interventions: Dietary Supplement: Postbiotic + nutritional recommendations
- Placebo group (Placebo Comparator): Gummy containing placebo formula.
  Interventions: Dietary Supplement: Placebo + nutritional recommendations

INTERVENTIONS:
Dietary Supplement: Postbiotic + nutritional recommendations — Study participants will consume daily one gummy containing a postbiotic formulation, along with adherence to healthy nutritional recommendations for 12 weeks.
  Arms: Postbiotic group
Dietary Supplement: Placebo + nutritional recommendations — Study participants will consume daily one gummy containing a placebo formulation, along with adherence to healthy nutritional recommendations for 12 weeks.
  Arms: Placebo group

SUMMARY:
The principal objective of this project is to evaluate the effect of a postbiotic supplement (inactivated microorganism) on body composition and other physiological and metabolic parameters related to excess body weight in overweight or obese adult men and women, as well as to determine changes in the gut microbiota associated with these outcomes.

Specific objectives are focus on evaluate the effect of the intervention on the following parameters:

* Changes in body weight and composition.
* Changes in glucose tolerance.
* Changes in gut microbiota (metagenomics).
* Changes in urinary and serum metabolites.
* Changes in routine biochemical variables related to carbohydrate and lipid metabolism, as well as liver parameters.
* Changes in specific markers involved in obesity pathology, such as insulin, leptin, adiponectin, and cytokines MCP-1, TNF, CRP, and others.
* Adherence to the nutritional recommendations and the gummy containing postbiotic formula.
* Changes in the level of physical activity.

Target sample size is 114 subjects, including a 10% of drop out.

Participants will be allocated in two groups for 12 weeks:

* Experimental group (n=57): nutritional recommendations + postbiotic supplement/gummy.
* Placebo group (n=57): nutritional recommendations + placebo supplement/gummy.

Participants will visit the nutritional intervention unit at weeks 1 and 12. A follow-up phone call will be conducted at week 6.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will complete an online questionnaire to verify eligibility based on the main inclusion criteria. Volunteers who meet these criteria will be invited to an information and screening visit to address any questions. Those who agree to participate will sign the informed consent form, be randomly assigned to one of the two study arms, and receive the necessary study materials.

During the intervention, volunteers will attend two clinical investigation visits. The Clinical Investigation Day 1 will be conducted on the first day of the study, and the Clinical Investigation Day 2 visit will occur at the end of the 12-week intervention. At both visits, anthropometric and body composition measurements, blood pressure, and samples of blood, urine, and stool will be collected. Additionally, data on diet, physical activity, sleep, and gastrointestinal symptoms will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 70 years.
* Volunteers with overweight or obesity (BMI: ≥ 27-39.9 kg/m²) and a body fat percentage of ≥ 30% for women and ≥ 20% for men.
* Stable body weight (±5%) for at least the three months prior to study initiation.
* Normal physical examination and vital signs, or clinically non-relevant findings for the purposes of the study (i.e., not related to metabolic health).
* Subjects must be able to understand and willing to sign the informed consent form, and comply with all study procedures and requirements.
* Continued pharmacological/hormonal treatment will be permitted provided it does not affect the study parameters and that the dosage has remained stable at least the previous three months to the start of the intervention. Treatment with insulin or any drug with a hypoglycemic effect will be excluded
* Willingness to undergo all study procedures (including the daily consumption of a 1 g gummy during the intervention).
* Time and geographic availability to attend the two on-site clinical evaluation sessions at the scheduled times (including a 3-hour session during visit 2).

Exclusion Criteria:

* Volunteers undergoing pharmacological treatment will be excluded if the treatment has not been stable for at least 3 months prior to study initiation. Excluded treatments include:
* Those that alter gastrointestinal function.
* Chronic use of stomach protectors.
* Any hypoglycemic drugs or insulin.
* Subjects with significant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, chronic reflux, etc.
* Subjects who have undergone surgical interventions resulting in permanent sequelae in the digestive tract (e.g., gastroduodenostomy) or bariatric surgery.
* Subjects with chronic metabolic diseases or obesity-related conditions, or systemic intestinal, hepatic, or renal diseases, including type 1 or 2 diabetes, severe dyslipidemia, uncontrolled thyroid disorders, cirrhosis, inflammatory bowel disease, untreated anemia, etc. (Non-alcoholic fatty liver disease will not be an exclusion criterion).
* Exceeding the alcohol consumption limit established for each sex (more than 14 units per week for women and 20 units per week for men).
* Pregnant or breastfeeding women, or those planning to become pregnant.
* Use of nutritional supplements (such as weight loss supplements, newly initiated fiber supplements, probiotics, postbiotics, etc.) containing compounds that may affect study outcomes, unless the participant agrees to discontinue them during the 12-week intervention period and a minimum 15-day washout period prior to baseline measurements is ensured.
* Blood donation within 14 days prior to the baseline visit.
* Subjects with any type of cancer or undergoing cancer treatment, or for whom less than 5 years have passed since remission.
* Subjects allergic to any component of the study product or to any other food that could interfere with or hinder study compliance.
* Subjects presenting any type of cognitive and/or psychiatric impairment.
* Subjects anticipated to have poor compliance or who, in the investigator's opinion, may have difficulty adhering to study procedures.
* Subjects currently undergoing treatment for weight loss or body composition modification.
* Subjects who are taking or have taken antibiotics within 60 days prior to the baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Body fat mass percentage | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body fat of participants will be analyzed by bioimpedance and reported in percentage and kilograms.

SECONDARY OUTCOMES:
Body weight | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body mass index will be calculated as follows: weight (kilograms)/ height (cm)2
Body lean mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body leen mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body water mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body water mass of participants will be analyzed by bioimpedance and reported in kilograms and percentage.
Body bone mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body bone mass of participants will be analyzed by bioimpedance and reported in kilograms.
Waist circumference | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Hip circumference | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Neck circumference | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Systolic blood pressure | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Diastolic blood pressure | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Heart rate | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in pulses/min.
Glucose concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Insulin concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood insulin concentration will be analyzed after an overnight fast by ELISA kit.
Blood glycated hemoglobin | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fasting blood glycated hemoglobin will be reported in percentage.
HOMA index | Clinical Investigation Day 1 and Clinical Investigation Day 2
  HOMA index will be calculated as follows: HOMA-IR = [fasting glucose (mmol/L) x fasting insulin (μU/ml)] / 22.5.
Total cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
HDL cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
LDL cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Triglyceride concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Aspartate aminotransferase | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Aspartate aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Alanine aminotransferase | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Alanine aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Gamma-glutamyl transferase | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Gamma-glutamyl transferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Leptine | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood leptine concentration will be analyzed after an overnight fast by ELISA kit.
Adiponectin | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood adiponectin concentration will be analyzed after an overnight fast by ELISA kit.
Monocyte Chemoattractant Protein-1 (MCP1) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood MCP1 concentration will be analyzed after an overnight fast by ELISA kit.
Tumor necrosis factor alpha (TNF-alpha) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood TNF-alpha concentration will be analyzed after an overnight fast by ELISA kit.
C Reactive protein (CRP) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood CRP concentration will be analyzed after an overnight fast by ELISA kit.
Albumin concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer.
Creatinine concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in μmol/L.
Life quality | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Life quality of participants will be evaluated by SF-36 questionnaire.
Gastrointestinal symptoms | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Physical activity | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Physical activity will be evaluated by the reduced version of the International Physical Activity Questionnaire, which estimates the total physical activity in MET-min/week, time spent sitting and classifies subjects based on their physical activity
Dietary intake | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Dietary intake (energy, macronutrients and micronutrients) will be analysed by food frequency questionnaire.
Chronotype | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Morningness-Eveningness Questionnaire (MEQ)
Depression | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Depression will be evaluated by Beck questionnaire.
Anxiety | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Anxiety will be evaluated by Stai questionnaire.
Lipidomic | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Lipidomic will be analyzed in plasma and serum.
Urine untargeted metabolomics | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Untargeted metabolomics will be analyzed in urine.
Blood untargeted metabolomics | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Untargeted metabolomics will be analyzed in plasma and serum.
Fecal microbiota | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fecal microbiota of participants will be analyzed by bacterial 16S or Shotgun gene sequencing technology.
Adherence to supplement consumption | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Adherence will be assessed using the supplement consumption record form.
Blood lipopolysaccharide (LPS) levels | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood LPS concentration will be analyzed by ELISA kit.
Blood zonulin levels | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Zonulin concentration will be analyzed by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Aranaz, PhD, Principal Investigator — Center for Nutrition Research; Fermín Milagro, PhD, Study Chair — Center for Nutrition Research; Idoia Ibero, PhD, Study Chair — Center for Nutrition Research; Blanca Martínez, Study Chair — Center for Nutrition Research; María Goñi, Study Chair — Center for Nutrition Research; Salomé Pérez, Study Chair — Center for Nutrition Research; Verónica Ciaurriz, Study Chair — Center for Nutrition Research; Ana Lorente, Study Chair — Center for Nutrition Research
Locations (1):
- Center for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No